CLINICAL TRIAL: NCT06467253
Title: Comparison of Two Non-invasive Neuromodulation Techniques as Synergistic Therapy to Cognitive Stimulation in Amnestic Mild Cognitive Impairment (aMCI): Genetic Characterization, Proteins Associated With Neurogenesis, Clinical, Neuroimaging and Electrophysiological Markers
Brief Title: Comparison of Two Non-invasive Neuromodulation Techniques as Synergistic Therapy to Cognitive Stimulation in Amnestic Mild Cognitive Impairment (aMCI)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Nacional de Psiquiatría Dr. Ramón de la Fuente (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IC20137.0
Record Dates: First submitted 2024-03-21; First posted 2024-06-20 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Mild Cognitive Impairment
Keywords: Mild cognitive impairment; Repetitive Transcranial Magnetic Stimulation rTMS; Transcranial Direct Current Stimulation tDCS; Neuromodulation Techniques; Amnestic Mild Cognitive Impairment; Cognitive Stimulation
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: Comparative, double-blind, randomized controlled clinical trial.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 1. rTMS + CS (Active Comparator): Repetitive Transcranial Magnetic Stimulation (rTMS) + Cognitive Stimulation (CS)
  Interventions: Device: 1. rTMS + CS
- 2. rTMS Sham + CS (Sham Comparator): Repetitive Transcranial Magnetic Stimulation Sham (rTMS Sham) + Cognitive Stimulation (CS)
  Interventions: Device: 2. rTMS Sham + CS
- 3. tDCS + CS (Active Comparator): Transcranial Direct Current Stimulation (tDCS) + Cognitive Stimulation (CS)
  Interventions: Device: 3. tDCS + CS
- 4. tDCS Sham + CS (Sham Comparator): Transcranial Direct Current Stimulation Sham (tDCS Sham) + Cognitive Stimulation (CS)
  Interventions: Device: 4. tDCS Sham + CS

INTERVENTIONS:
Device: 1. rTMS + CS — In the first phase each participant will receive 15 sessions of rTMS and 9 sessions of CS divided in 3 weeks, in the maintenance phase each participant will receive 1 session of rTMS and 1 session of CS per week for 12 weeks. Each session will consist of 10 trains of 10 stimuli, at a 5-Hz frequency and a stimulation intensity of 120% of the resting motor threshold.
  rTMS will be administered by a MagPro R30 stimulator (MagVenture) and an active/placebo 8-shape coil model MCF-B70.
  Two surface electrodes will be employed to replicate rTMS skin sensations near the stimulation site. The rTMS condition will be double-blinded through the use of a USB stick.
  Cognitive stimulation will be a Mexican adaptation of the "Memory Training and Cognitive Stimulation for Mild Cognitive Impairment" from the Center for the Prevention of Cognitive Impairment of the Madrid City Council.
  In total, each participant will receive 27 sessions of rTMS and 21 sessions of CS.
  Arms: 1. rTMS + CS
Device: 2. rTMS Sham + CS — In the first phase each participant will receive 15 sessions of rTMS Sham and 9 sessions of CS divided in 3 weeks, in the maintenance phase each participant will receive 1 session of Sham rTMS and 1 session of CS per week for 12 weeks.
  In total, each participant will receive 27 sessions of Sham rTMS and 21 sessions of CS.
  rTMS will be administered by a MagPro R30 stimulator (MagVenture) and an active/placebo 8-shape coil model MCF-B70.
  Two surface electrodes will be employed to replicate rTMS skin sensations near the stimulation site. The sham condition will be double-blinded through the use of a USB stick.
  Cognitive stimulation will be a Mexican adaptation of the "Memory Training and Cognitive Stimulation for Mild Cognitive Impairment" from the Center for the Prevention of Cognitive Impairment of the Madrid City Council.
  In total, each participant will receive 27 sessions of rTMS and 21 sessions of CS.
  Arms: 2. rTMS Sham + CS
Device: 3. tDCS + CS — In the first phase each participant will receive 15 sessions of tDCS and 9 sessions of CS divided in 3 weeks, in the maintenance phase each participant will receive 1 session of tDCS and 1 session of CS per week for 12 weeks. Each session will consist of the delivery of a weak direct current of 2mA for 30 minutes.
  tDCS will be administered by the Sooma tDCS stimulator. The tDCS condition will be double-blinded, and a third operator will program the stimulator.
  Cognitive stimulation will be a Mexican adaptation of the "Memory Training and Cognitive Stimulation for Mild Cognitive Impairment" from the Center for the Prevention of Cognitive Impairment of the Madrid City Council.
  In total, each participant will receive 27 sessions of tCDS and 21 sessions of CS.
  Arms: 3. tDCS + CS
Device: 4. tDCS Sham + CS — In the first phase each participant will receive 15 sessions of tDCS Sham and 9 sessions of CS divided in 3 weeks, in the maintenance phase each participant will receive 1 session of Sham tDCS and 1 session of CS per week for 12 weeks.
  tDCS will be administered by the Sooma tDCS stimulator. The sham condition will be double-blinded, and a third operator will program the stimulator.
  Cognitive stimulation will be a Mexican adaptation of the "Memory Training and Cognitive Stimulation for Mild Cognitive Impairment" from the Center for the Prevention of Cognitive Impairment of the Madrid City Council.
  In total, each participant will receive 27 sessions of Sham tDCS and 21 sessions of CS.
  Arms: 4. tDCS Sham + CS

SUMMARY:
This is a comparative, double-blind, randomized controlled clinical trial for people with Amnestic Mild Cognitive Impairment. The investigators will compare the effects of two non-invasive neuromodulation techniques (Repetitive Transcranial Magnetic Stimulation and Transcranial Direct Current Stimulation) combined with cognitive stimulation. These non-invasive neuromodulating techniques will be applied as a treatment alternative to be able to compare non-invasive techniques with cognitive stimulation CS alone, taking into account clinical and neuropsychological evaluations in addition to: 1) the known clinical risk factors (physical activity, comorbidities treatment, etc.) that allow the investigators to characterize the participants; 2) characterize the participants with genetic biomarkers using the APOE4, CR1, COMT, TREM2 and ABCA7 genotype; 3) document the biological effects related to neurogenesis from olfactory epithelial neural progenitor cells and solubles factors of serum; 4) use hippocampal volume, cortical thickness of the medial temporal cortex and parietal cortex by means of structural magnetic resonance imaging and the default mode network by means of functional magnetic resonance imaging at rest as a biomarker of response to treatment and 5) associate the response to treatment with changes in Motor Evoked Potential (MEP) amplitude and latency in order to generate a response-to-treatment biomarker with neuromodulators in Mild Cognitive Impairment (MCI) and changes in electroencephalogram.

DETAILED DESCRIPTION:
Mild Cognitive Impairment can be described as an intermediate stage between intact cognition and dementia, this study has become a global priority due to alarming changes in the population pyramid that place the world population at a higher risk of developing dementia. The global prevalence of MCI is between 15-20% in people over 60 years old. In 2012, a prevalence of MCI of 3.2% was found in Mexico City, which encourages the researchers to study this phenomenon to achieve early detection and create interventions that could delay the onset of dementia and even prevent it. Symptomatology is distinguished by deficits in one or more cognitive domains through formal tests applied repeatedly; the individual can manifest symptoms directly by identifying as different from a previous state and/or being corroborated by an informant. The amnestic cognitive impairment (aMCI) occurs when the cognitive failure is limited only to the domain of episodic memory. Generally, there is a slight functional impairment for complex tasks, but the basic and instrumental activities of daily life must be preserved. Behavioral and psychological symptoms (BPSD) can occur. Apathy, anxiety, and depression present in patients with mild cognitive impairment may represent an increased risk of dementia and in many cases, can be the first symptoms to appear. The evaluation is essential because BPSD are often controllable with treatment and appears in up to 77% of patients with MCI.

Despite the need to stop the progression to dementia, a MCI treatment is currently nonspecific, focused on associated events, with pharmacological and non-pharmacological measures aimed to reduce cognitive and neuropsychiatric symptoms. Therapeutic methods that promote neuroplasticity, for instance, cognitive stimulation (CS) and non-invasive neuromodulatory techniques such as Repetitive Transcranial Magnetic Stimulation (rTMS) and Transcranial Direct Current Stimulation (tDCS), optimize performance by stimulating the neural network distributed around a dysfunctional circuit, interacting with brain plasticity, and inducing or increasing compensatory mechanisms. This phenomenon could add to the cognitive reserve and interfere with the temporal evolution of the symptoms. Thereby, the rTMS and tDCS have been suggested as a possible treatment in aMCI. These non-invasive alternatives (rTMS and tDCS) have shown efficacy as a treatment in other disorders, but evidence is required on the efficacy, tolerability, and viability of the application in patients with amnesic MCI as well as the time that the effect of its application remains, which creates the need of further studies with maintenance phases.

In this project, the researchers propose a clinical trial for participants with risk of developing dementia using rTMS and tDCS added to CS in an effectiveness comparison using strict placebo control methods which will only be used with rTMS and tDCS, not with CS. The non-invasive neuromodulating techniques will be applied as a treatment alternative to be able to compare the techniques with CS alone, taking into account clinical and neuropsychological evaluations in addition to: 1) the known clinical risk factors (physical activity, comorbidities treatment, etc.) that allow to characterize patients; 2) characterize the participants with genetic biomarkers using the APOE4, CR1, COMT, TREM2 and ABCA7 genotype; 3) document the biological effects related to neurogenesis from olfactory epithelial neural progenitor cells isolated before and after treatment. In addition to the documentation of soluble factors secreted by olfactory epithelial neural progenitor cells, what is relevant to the knowledge of the influence of peripheral serum on microglia. This is crucial role in inflammation. The evaluations will be performed at different time points such as: Baseline (T0), after first phase of treatment (T1=15 sessions/week of tDCS+CS), after maintenance (T2=12 sessions/week of tDCS+CS), and follow-up phase (T3=1 year after treatment); 4) use hippocampal volume, cortical thickness of the medial temporal cortex and parietal cortex using structural magnetic resonance imaging and the default mode network using functional magnetic resonance imaging at rest as a biomarker of response to treatment and 5) associate the response to treatment with changes in Motor Evoked Potential (MEP) amplitude to generate a response-to-treatment biomarker with neuromodulators in MCI and changes in electroencephalogram (EEG).

Among the current limitations on knowledge of this disease, many studies use biomarkers to predict MCI or progression to dementia, and although most biomarkers are reported to be valuable in this setting, few are compared with each other, so this is currently difficult to understand the relative importance of the different biomarkers when used together. For this reason, the present project could be a contribution in the short and long term to detect changes that may or may not be related to each other and generate multiple lines of research.

Population aging will continue to increase and therefore there will be a greater number of people with aMCI. Currently, there is no treatment that prevents the progression of aMCI to AD, so the trend is to make earlier interventions. aMCI is a condition of opportunity because the cognitive reserve of the patients has not been exhausted, so developing studies with innovative treatments and few side effects that can change the evolution over time is important. To that end, understanding the etiology of this progression and designig treatments that delay or definitively stop aMCI are of importance to preserve the functionality of individuals with this condition.

Clinical trials with rTMS and tDCS carried out in aMCI have already shown favorable results regarding episodic memory, semantic memory, and speed of information processing. This trial will be able to contribute to the already reported findings that allow to identify better therapeutic approaches that support the standardization of the application of neuromodulatory techniques. Besides, the possible additive effect of neuromodulatory techniques and CS is well known, but no studies are comparing between diferent interventions with each other. The genetic characterization will be obtained, an experimental biomarker of secretion proteins from olfactory epithelial neural progenitor cells together with the analysis of the neurogenic process occurring in the olfactory epithelium will be generated, an experimental biomarker of serum and the effects soluble factors contained in serum on microglia will be generated, neuroimaging and produce neurophysiological measures considered as possible neuroplasticity biomarkers (MEPs and EEG) associated with the response to non-pharmacological treatment will be recorded and evaluated if the parameters are related to clinical and cognitive characteristics. With this therapeutic approach where non-invasive neuromodulatory techniques are combined with CS, the aim is to improve the quality of care for patients with aMCI, considering that neuromodulation alternatives can delay the process of deterioration in each patient admitted.

The hypotheses in this study are: 1) The combined application of non-invasive neuromodulation techniques with cognitive stimulation will significantly improve the cognitive performance of patients with aMCI, compared to the single application of non-invasive neuromodulation techniques or cognitive stimulation alone. 2) There will be differences in the protein expression in the olfactory epithelial neural progenitor cells of patients with aMCI who are treated with some non-invasive neuromodulation techniques and those who only receive cognitive stimulation. 3) The soluble factors in the serum of patients with aMCI before and after treatment will differentially modulate microglia. 4) There will be differences in brain morphology such as cortical thickness and surface area, white matter integrity, as well as structural connectivity between different brain areas before and after treatment with non-invasive stimulation techniques. 5) There will be differences in the amplitude and latency of the MEP as well as changes in EEG of patients with aMCI who are treated with one of the non-invasive neuromodulation techniques and patients who only receive CS.

ELIGIBILITY:
Inclusion criteria:

* Being vaccinated against the SARS-COV2 virus.
* Speak Spanish fluently.
* Level of schooling greater than or equal to 6 years.
* Amnestic mild cognitive impairment established by clinical examination performed by the treating physician (MoCA score: 19-25 points for probable aMCI) (based on the National Institute on Aging and Alzheimer's Association (NIA/AA) criteria, 2011).
* Adequate visual and auditory acuity to perform neuropsychological tests and cognitive rehabilitation.
* If receiving psychotropic drugs, having started the drugs at least 12 weeks before the start of the study, remaining at stable doses, or having suspended the drugs for at least 4 weeks before the study.
* Be in good health without non-psychiatric medical diseases (uncontrolled systemic arterial hypertension, diabetes mellitus or dyslipidemia, infections, thyroid disease, vitamin deficiency) interfering with the study.
* Willingness to participate in a study scheduled for 8 weeks and that participants can go to the Instituto Nacional De Psiquiatría for treatments, as well as scheduled evaluations.
* An informant to respond to some of the assessment questionnaires throughout the study and who would stay with the participant for at least 10 h/week.

Exclusion Criteria:

* Any neurological disease that raises suspicion of cognitive failure other than Alzheimer's disease, such as Parkinson's, multi-infarct dementia, Huntington's disease, hydrocephalus, brain tumor, progressive supranuclear palsy, seizure disorder, subdural hematoma, multiple sclerosis, history of trauma craniocerebral with loss of alertness.
* Participants with a history of severe psychiatric disorders according to DSM-5 (bipolar disorder, schizophrenia, chronic depression) or with psychotic features, agitation, or behavioral problems in the last three months that could lead to difficulties in meeting the protocol.
* History of psychoactive substance abuse and current alcohol consumption with a pattern of abuse or dependence in the last two years.
* Participants with alterations in a conventional electroencephalogram (paroxysmal phenomena identified by a neurophysiologist).
* Participants with pacemakers, intracranial metal objects, or history of brain surgery, aneurysm clips, artificial heart valves, ear implants, metal fragments, or foreign objects in the eyes, skin, or body.
* Participation in the last 6 months in a clinical study that involved neuropsychological assessment.

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-06-15 (Estimated)

PRIMARY OUTCOMES:
Changes in orientation | Baseline, after maintenance (15 weeks), and in follow-up phase (1 year later).
  Measured by the Barcelona Test. Score ranges from 10 or less to 95. Direct scores are converted to percentile. Higher scores mean better outcomes.
Changes in language | Baseline, after maintenance (15 weeks), and in follow-up phase (1 year later).
  Measured by the WAIS-IV vocabulary test. Score ranges from 1 to 19. Direct scores are converted to standardized scores. Higher scores mean better outcomes.
Changes in language | Baseline, after maintenance (15 weeks), and in follow-up phase (1 year later).
  Measured by the Barcelona Test. Score ranges from 10 or less to 95. Direct scores are converted to percentile. Higher scores mean better outcomes.
Changes in verbal memory | Baseline, after maintenance (15 weeks), and in follow-up phase (1 year later).
  Measured by the Barcelona Test. Score ranges from 10 or less to 95. Direct scores are converted to percentile. Higher scores mean better outcomes.
Changes in verbal memory | Baseline, after maintenance (15 weeks), and in follow-up phase (1 year later).
  Measured by Neuropsi Attention and Memory. Score ranges from 1 to 19. Direct scores are converted to standardized scores. Higher scores mean better outcomes.
Changes in visual memory | Baseline, after maintenance (15 weeks), and in follow-up phase (1 year later).
  Measured by the Barcelona Test. Score ranges from 10 or less to 95. Direct scores are converted to percentile. Higher scores mean better outcomes.
Changes in visual memory | Baseline, after maintenance (15 weeks), and in follow-up phase (1 year later).
  Measured by Neuropsi Attention and Memory. Score ranges from 1 to 19. Direct scores are converted to standardized scores. Higher scores mean better outcomes.
Changes in visual-constructive abilities | Baseline, after maintenance (15 weeks), and in follow-up phase (1 year later).
  Measured by the Barcelona Test. Score ranges from 10 or less to 95. Direct scores are converted to percentile. Higher scores mean better outcomes.
Changes in visual-constructive abilities | Baseline, after maintenance (15 weeks), and in follow-up phase (1 year later).
  Measured by Neuropsi Attention and Memory. Score ranges from 10 or less to 95. Direct scores are converted to standardized scores. Higher scores mean better outcomes.
Changes in processing speed | Baseline, after maintenance (15 weeks), and in follow-up phase (1 year later).
  Measured by the Barcelona Test. Score ranges from 10 or less to 95. Direct scores are converted to percentile. Higher scores mean better outcomes.
Changes in processing speed | Baseline, after maintenance (15 weeks), and in follow-up phase (1 year later).
  Measured by the Trail Making Test version A and B. Score ranges from 5 to 95. Direct scores are converted to percentile. Higher scores mean better outcomes.
Changes in abstraction | Baseline, after maintenance (15 weeks), and in follow-up phase (1 year later).
  Measured by the Barcelona Test. Score ranges from 10 or less to 95. Direct scores are converted to percentile. Higher scores mean better outcomes.
Changes in verbal fluency | Baseline, after maintenance (15 weeks), and in follow-up phase (1 year later).
  Measured by a verbal fluency test (semantic: animals and phonologic: F, A, S). Score ranges from 5 to 95. Direct scores are converted to percentile. Higher scores mean better outcomes.
Changes in interference | Baseline, after maintenance (15 weeks), and in follow-up phase (1 year later).
  Measured by the Stroop Test. Score ranges from 5 to 95. Direct scores are converted to percentile. Higher scores mean better outcomes.
Changes in working memory | Baseline, after maintenance (15 weeks), and in follow-up phase (1 year later).
  Measured by the Barcelona Test. Score ranges from 10 or less to 95. Direct scores are converted to percentile. Higher scores mean better outcomes.
Changes in working memory | Baseline, after maintenance (15 weeks), and in follow-up phase (1 year later).
  Measured by Trail Making Test version A and B. Score ranges from 5 to 95. Direct scores are converted to percentile. Higher scores mean better outcomes.
Changes in Global Cognitive Function | Baseline, after first phase (3 weeks), after maintenance (15 weeks) and in follow-up phase (1 year later).
  Measured by Montreal Cognitive Assessment. Score ranges from 0 to 30 points. Higher scores mean better outcomes.
Changes in Global Cognitive Function | Baseline, after first phase (3 weeks), after maintenance (15 weeks) and in follow-up phase (1 year later).
  Measured by Screen for Cognitive Impairment in Psychiatry. Direct scores ranges from 37 to 115 points. Higher scores mean better outcomes.
Changes in memory regarding situations and activities of daily life | Baseline, after first phase (3 weeks), after maintenance (15 weeks) and in follow-up phase (1 year later)
  Measure by Everyday Memory Questionnaire. Score ranges from 0 to 56. Higher scores mean worse outcomes.
Changes in Global Clinical Impression | Baseline, after first phase (3 weeks), after maintenance (15 weeks) and in follow-up phase (1 year later).
  Measure by Clinical Impression Scale. Score ranges from 0 to 7. Higher scores mean worse outcomes.
Changes in Motor Evoked Potentials | Baseline, after first phase (3 weeks), after maintenance (15 weeks) and in follow-up phase (1 year later).
  Measured by MagVenture, Transcranial Magnetic Stimulation (TMS). Evaluation of cortical excitability and synaptic plasticity using a 5 Hz-rMTS (repetitive TMS). Increased amplitude and decreased latency parameters mean better outcomes after the intervention.
Changes in Olfactory Epithelial Neural Progenitor Cells | Baseline, after first phase (3 weeks), after maintenance (15 weeks) and in follow-up phase (1 year later).
  Measured by Neural Progenitor Cells Isolated. Quantification of the number of neural progenitor cells isolated from the olfactory epithelium. Increased number of neural progenitor cells after the intervention.
Changes in Solubles Factors of Serum | Baseline, after first phase (3 weeks), after maintenance (15 weeks) and in follow-up phase (1 year later).
  Measured by Exosome Analysis.To find a differential content of inflammatory markers in the exosomes before and after the intervention.
Changes in Functional Magnetic Resonance Imaging | Baseline, after first phase (3 weeks), after maintenance (15 weeks) and in follow-up phase (1 year later).
  Measured by Philips Magnetic Resonator, Ingenia 3T Equipment. The Sternberg task, which stimulates working memory and recent memory, will be used to observe changes Bold signal changes in gray matter, the hippocampus and white matter tracts.

SECONDARY OUTCOMES:
Changes in Apathy symptoms | Baseline, after first phase (3 weeks), after maintenance (15 weeks) and in follow-up phase (1 year later).
  Measured by Apathy Evaluation Scale (self-report, informant report and clinician report). Score ranges from 18 to 72. Higher scores mean worse outcomes.
Changes in Depression | Baseline, after first phase (3 weeks), after maintenance (15 weeks) and in follow-up phase (1 year later).
  Measured by Yesavage Geriatric Depression Scale. Score ranges from 0 to 30. Higher scores mean worse outcomes.
Changes in behavioral and psychological symptoms | Baseline, after first phase (3 weeks), after maintenance (15 weeks) and in follow-up phase (1 year later).
  Measured by Cummings Neuropsychiatric Inventory. Score ranges for frequency are 1 to 4, severity score ranges from 1 to 3 and distress score ranges from 0 to 4. Higher scores mean worse outcomes.
Changes in electroencephalogram | Baseline, after first phase (3 weeks), after maintenance (15 weeks) and in follow-up phase (1 year later).
  Measured in each frequency band (delta, theta, alfa beta y gamma) before and after the intervention with the small-worldness measure, which will be obtained in order to observe the global optimization in the transmission of brain information. Likewise, will be complemented with an analysis of the clustering coefficient, local efficiency and global efficiency, calculating these measures in the F3 and F4 regions. To find changes in the small-worldness after the intervention.
Changes in smell identification | Baseline, after first phase (3 weeks), after maintenance (15 weeks) and in follow-up phase (1 year later).
  Measured by the Brief Smell Identification Test. Score ranges from 0 to 12. Higher scores mean better outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Ruth Alcalá Lozano, Dr., Principal Investigator — Instituto Nacional de Psiquiatría Ramón de la Fuente Muñiz
Locations (1):
- Instituto Nacional de Psiquiatría Ramón de la Fuente Muñiz, Mexico City, Mexico